CLINICAL TRIAL: NCT06205004
Title: Prevalence of Internet Addiction and it's Effects on Psychological Well-being of Adults in Hong Kong
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Other Study IDs: Prevalence of IA in Adults
Record Dates: First submitted 2023-11-20; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-11

CONDITIONS: Internet Addiction
Keywords: Internet Addiction; Quality of life; Young Adults
MeSH Terms: conditions — Internet Addiction Disorder | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young adults in HK: questionnaire based study
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — In the present study, the investigators aim to investigate the prevalence and effects of IA on the psychosocial well-being among adults in Hong Kong by measuring the level of Internet use, depression, anxiety, sleep quality, QOL together with basic demographic data in the current situation of COVID with popularity of Metaverse.

SUMMARY:
The goal of this quantitative study is to learn about the the prevalence of internet addiction and its effects on psychological well-being of adults in Hong Kong. The main question it aims to answer is:

• What is the prevalence of internet addiction and its effects on psychological well-being of adults in Hong Kong

Participants will be invited to complete a set of questionnaire that includes assessment on their level of Internet use, depression, anxiety, sleep quality, QOL together with basic demographic data in the current situation of COVID with popularity of Metaverse..

DETAILED DESCRIPTION:
Internet addiction (IA) appeared to become serious issues since the emergence of Internet over the decades. The definition of Internet Penetration Rate (IPR) is the percentage of the entire population who has Internet usage. As of July 2022, Denmark, the UAE, and Ireland had the highest IPR, all recording 99% of their population accessing the internet. While in Hong Kong, it has reached 93.6%, not far from the first in Asia - South Korea (98%). The widespread use has shown the popularity of Internet is skyrocketing through the years.

Despite there are several studies conducted on IA from the West, the results might not be not applicable in adults in Hong Kong due to various reasons such as policies against COVID and cultural difference as lifestyle, living and social environment, family relationship style. Those might have potential influence on the engagement in physical and social activities and involvement in Internet. In addition to the emergence of Metaverse, situations, policies and people's attitude towards COVID might have changed drastically and affect the prevalence of IA in Hong Kong adult. To conclude, the effect of COVID and Metaverse on the prevalence of IA in adults in Hong Kong and the mechanisms/reasons behind is unclear.

In the present study, the investigators aim to investigate the prevalence and effects of IA on the psychosocial well-being among adults in Hong Kong by measuring the level of Internet use, depression, anxiety, sleep quality, QOL together with basic demographic data in the current situation of COVID with popularity of Metaverse.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-40
* Resided in Hong Kong
* Can speak Cantonese and write Chinese

Exclusion Criteria:

* Self-reported to have identified cognitive problems and communication problems

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In terms of population size, in Hong Kong, young adults occupied 26.4%-28.2% among the total population, which comparatively appeared to be a greater group than adolescents aged from 13 to 17 (3.8%). Moreover, as fertility and birth rate in Hong Kong continued to shrank to lowerst in 56 years due to multiple factors, it is estimated that the
  whole population is aging and adults would be the main population in these few decades. Besides, according to the Labour Force Census, as at 2021, the highest labour force participation rate falls in age group of 25-44. Being a large population and labour force in Hong Kong, the IA behaviour of young adults are crucial to maintain productivity and social functioning. Hence this study will focus on studying young adults.
Sampling Method: Probability Sample
Enrollment: 298 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
prevalence of Internet Addiction | at day 1
  Internet Addiction Test (IAT-20) developed by Young, 1998

SECONDARY OUTCOMES:
Overall Quality of Life | at day 1
  Short-Form Six-Dimension (SF-6D) by Professor John Brazier and Jennifer Roberts
Depression | at day 1
  Center for Epidemiologic Studes Depression scale (CES-D) by Radloff, 1977
Anxiety | at day 1
  Generalized Anxiety Disorder-7 (GAD-7) by Spitzer et al, 2006
Sleep Quality | at day 1
  The Pittsburgh Sleep Quality Index (PSQI) by Buysse et al, 1989

CONTACTS AND LOCATIONS:
Locations (1):
- Katherine Lam, Hong Kong, Hong Kong,China, Hong Kong

IPD SHARING:
Plan to Share IPD: No
All personal data will only be accessable within the research team, for research purpose.